CLINICAL TRIAL: NCT02194205
Title: A One-year Randomized, Double-blind, Placebo and Active-controlled Parallel Design Safety and Efficacy Comparison of COMBIVENT HFA Inhalation Aerosol to COMBIVENT (CFC) Inhalation Aerosol in Patients With COPD
Brief Title: Comparison of Safety and Efficacy of COMBIVENT HFA to COMBIVENT (CFC) in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1012.11
Record Dates: First submitted 2014-07-17; First posted 2014-07-18 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (4):
- COMBIVENT HFA (Experimental)
  Interventions: Drug: COMBIVENT HFA
- Placebo HFA (Placebo Comparator)
  Interventions: Drug: Placebo HFA
- COMBIVENT (CFC) (Active Comparator)
  Interventions: Drug: COMBIVENT CFC
- Placebo CFC (Placebo Comparator)
  Interventions: Drug: Placebo CFC

INTERVENTIONS:
Drug: COMBIVENT HFA
  Arms: COMBIVENT HFA
Drug: Placebo HFA
  Arms: Placebo HFA
Drug: COMBIVENT CFC
  Arms: COMBIVENT (CFC)
Drug: Placebo CFC
  Arms: Placebo CFC

SUMMARY:
To compare the long-term (one-year) bronchodilator efficacy and safety of COMBIVENT hydrofluoroalkane (HFA) Inhalation Aerosol to COMBIVENT chlorofluorocarbon (CFC) Inhalation Aerosol and Placebo formulations of each in patients with COPD. In addition, steady state pharmacokinetics over one dosing interval following four weeks of therapy will be characterized.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of COPD
* Male or female patients 40 years of age or older
* Patients must have a smoking history of more than ten pack-years. A pack-year is defined as the equivalent of smoking one pack of 20 cigarettes per day for a year
* Patients must be able to perform technically satisfactory pulmonary function tests
* Patients must be able to be trained in the proper use of a metered dose inhalator (MDI)
* All patients must sign an Informed Consent Form prior to participation in the trial i.e. prior to pre-study washout of their usual pulmonary medications
* Patients must be on at least one regular aerosol bronchodilator for control of their COPD symptoms and have symptoms of bronchospasm (wheeze or shortness of breath) present OR Patients must be on at least two classes of prescribed bronchodilators on a regular basis for control of their COPD symptoms for the three month period immediately preceding the screening visit.

Exclusion Criteria:

* Patients with significant disease other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study
* Patients with clinically relevant abnormal baseline hematology, blood chemistry or urinalysis. If the abnormality defines a disease listed as an exclusion criterion, the patient is excluded
* All patients with a serum aspartate amino transferase (ASAT/SGOT) > 80 IU/L, serum alanine amino transferase (ALAT/SGPT) > 80 IU/L, bilirubin > 2.0 mg/dL or creatinine > 2.0 mg/dL will be excluded regardless of the clinical condition. Repeat laboratory evaluation will not be conducted in these patients.
* Patients who have a total bood eosinophil count >= 600 mm**3. A repeat eosinophil count will not be conducted in these patients
* Patients with a recent history (i.e. one year or less) of myocardial infarction
* Patients with a recent history (i.e. three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy
* Patients with a history of cancer, other than treated basal cell carcinoma, within the last five years
* Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis
* Patients who have undergone thoracotomy with pulmonary resection. Patients wth a history of thoracotomy for other reasons should be evaluated as per exclusion criterion No. 1
* Patients with a history of asthma, allergic rhinitis or atopy.
* Patients with a history of or active alcohol or drug abuse
* Patients with known active tuberculosis
* Patients with an upper respiratory tract infection or COPD exacerbation in the six weeks prior to the Screening Visit (Visit 1) or during the baseline period
* Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction
* Patients with known narrow-angle glaucoma
* Patients with current significant psychiatric disorders
* Patients with regular use of daytime oxygen therapy
* Patients who are being treated with beta-blocker medications, monoamine oxidase (MAO) inhibitors or tricyclic antidepressants
* Patients who are being treated with cromolyn sodium or nedocromil sodium
* Patients who are being treated with antihistamines
* Patients using oral corticosteroid medication at unstable doses or at a dose in excess of the equivalent of 10 mg of prednisone per day or 20 mg every other day
* Patients who have been treated with oral beta-adrenergics or long-acting beta-adrenergics in the two weeks prior to the Screening Visit or during the baseline period
* Patients who have had changes in their therapeutic plan within the last six weeks prior to the Screening Visit or during the baseline period, excluding changes from long acting or oral beta-adrenergics to short acting inhaled beta-adrenergics for purposes of this trial
* Pregnant of nursing women or woman of childbearing potential not using a medically approved means of contraception
* Patients with known hypersensitivity to anticholinergic or beta-agonist drugs or any other component of either COMBIVENT formulation
* Patients who have taken an investigational drug within one month or six half lives (whichever is greater) prior to Screening visit
* Previous participation in this study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2000-10; Primary Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
Area under the curve from 0 to 6 hours (AUC0-6) of forced expiratory volume in the first second (FEV1) | after 12 weeks

SECONDARY OUTCOMES:
Peak FEV1 response | 28 weeks
Onset of therapeutic FEV1 response | 28 weeks
Duration of therapeutic FEV1 response | 28 weeks
Time to peak FEV1 response | 28 weeks
Average FEV1 response as area under the curve from 0 - 6 hours divided by six (TAUC0-6) | 28 weeks
Average forced vital capacity (FVC) response area under the curve from 0 - 6 hours divided by six (AUC0-6) | 28 weeks
Number of participants requiring test-day rescue therapy | 28 weeks
Peak expiratory flow rate (PEFR) | 28 weeks
Daily COPD symptom scores | 28 weeks
Number of puffs of rescue medication | 28 weeks
Number and length of COPD exacerbations | 28 weeks
Average FEV1 response as area under the curve from 0 - 8 hours divided by six (TAUC0-8) | 28 weeks
Number of adverse events including paradoxical bronchoconstrictions | 28 weeks
Number of patients with clinically significant changes in pulse rate and blood pressure | 28 weeks
Plasma ipratropium concentration | pre-treatment, 5, 15, 30 min; 1, 2, 4 and 8 hours
Plasma albuterol concentration | pre-treatment, 5, 15, 30 min; 1, 2, 4 and 8 hours
Renal excretion of ipratropium fractions | pre-treatment, 0 - 2 hours, 2 - 8 hours
Renal excretion of albuterol fractions | pre-treatment, 0 - 2 hours, 2 - 8 hours
Physician's global evaluation on an 8-point scale | 28 weeks
Peak FVC response | 28 weeks
Number of patients with clinically significant changes in laboratory tests | 28 weeks
Number of patients with abnormal findings in physical examination | 28 weeks
Number of patients with clinically significant changes in electrocardiogram | 28 weeks